CLINICAL TRIAL: NCT00213824
Title: A Study of the Expression of Nogo and Reticulon Genes in Skeletal Muscle of Patients With Amyotrophic Lateral Sclerosis
Status: Terminated | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 3142
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; Nogo gene; reticulon genes
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — tissue (skeletal muscle)

SUMMARY:
This is a study of the expression of nogo and reticulon genes in the skeletal muscle of patients with amyotrophic lateral sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with definite ALS
* Males or females
* Age > 18

Exclusion Criteria:

* Patients with other neuromuscular affections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University Hospital, Strasbourg, France
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2004-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yon-Andoni Echaniz-Laguna, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (1):
- Clinique Neurologique, Service des Maladies du Système Nerveux et du Muscle, Hôpital Civil, Hôpitaux Universitaires, Strasbourg, France